CLINICAL TRIAL: NCT02963090
Title: A Randomized Phase II Study Evaluating Pembrolizumab vs Topotecan in the Second-Line Treatment of Patients With Small Cell Lung Cancer
Brief Title: Pembrolizumab vs Topotecan in Patients With Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AFT-17
Record Dates: First submitted 2016-10-26; First posted 2016-11-15 (Estimated); Results first posted 2022-09-16 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; small cell lung cancer; lung cancer; topotecan; pembrolizumab
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Topotecan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topotecan (Active Comparator): Topotecan IV at 1265mg/m^2 Days 1-5 of every 21 day cycle
  Interventions: Drug: Topotecan; Drug: Pembrolizumab
- Pembrolizumab (Experimental): Pembrolizumab IV 200mg infusion Day 1 of every 21 day cycle
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Topotecan — Topotecan at 1.25mg/m2 on days 1 to 5 every 21-days until progression of disease or unacceptable toxicities.
  Patients with progression of disease by RECIST 1.1 will be allowed cross over to receive pembrolizumab 200 mg IV every 21-days for up to 1 year until progression of disease or unacceptable toxicities.
  Other Names: hycamtin
  Arms: Topotecan
Drug: Pembrolizumab — 200 mg IV every 21-days until progression of disease or unacceptable toxicities.
  Other Names: Keytruda; MK-3475

SUMMARY:
This is a multi-institutional, randomized, open-label phase II study of pembrolizumab compared to topotecan, administered to patients with SCLC who have progressed or relapsed after first-line treatment with etoposide and platinum. Patients will be randomized in a 2:1 fashion to receive pembrolizumab or topotecan. Participants in the topotecan arm that progress will be allowed to cross-over to the pembrolizumab arm.

DETAILED DESCRIPTION:
Patients who meet the eligibility criteria and are randomized to one of the treatment arms, will receive either topotecan alone intravenously at 1.25 mg/m2 on days 1 to 5 of a 21-day cycle or pembrolizumab alone administered intravenously at 200mg every 21 days.

During the study period, patients will be evaluated clinically by physical exam and with routine blood work every 21 days. Adverse events will be monitored throughout the trial and graded in severity according to the guidelines outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4. Pre-specified adverse events of clinical interest include: 1) Grade ≥ 2 diarrhea, 2) Grade ≥ 2 colitis, 3) Grade ≥ 2 pneumonitis, 4) Grade ≥ 2 hepatitis 5) Grade ≥ 3 hypo- or hyperthyroidism.

Patients will be evaluated every 6 weeks (42 ± 7 days) with radiographic imaging to assess response to treatment. Investigators will make all treatment-based decisions using RECIST 1.1. Patients will continue to receive topotecan or pembrolizumab every three weeks until documented disease progression, unacceptable side effects, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the patient, patient withdraws consent, pregnancy of the patient, non-compliance with trial treatment or procedure requirements or administrative reasons. Patients on the topotecan arm who progress on study will be allowed to cross-over to the pembrolizumab arm.

After the end of treatment, each patient will be followed for a minimum of 30 days for adverse event monitoring. Serious adverse events will be collected for up to 90 days after the end of treatment or 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier. Immune related serious adverse events will be followed for 90 days after end of treatment. Subjects who discontinue treatment for reasons other than disease progression will have posttreatment follow-up every 6 weeks for disease status until progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone contact every 3 months for overall survival until death or withdrawal of consent.

Although subjects will be enrolled regardless of PD-L1 status, subjects will be required to provide tissue of a tumor lesion (either archived tissue or a new biopsy before initiating therapy). Tumor samples will be required before initiating therapy (preferably a new specimen) and a repeat biopsy will be performed, if clinically feasible, on-treatment (during weeks 4 to 6) for those in the pembrolizumab arm and at the time of disease progression for those in the topotecan arm. PD-L1 expression status by immunohistochemistry will be determined on tumors at baseline, on treatment and at the time of topotecan progression. Numerous other correlative studies also will be performed, as outlined below. Peripheral blood mononuclear cell samples will be collected at screening, at day 1 of cycles 1, 2 and 3, and at the time of each imaging study (while on study), for characterization of T-cell phenotypes to understand how changes may correlate with clinical response.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the patient must:

1. Have histologically or cytologically confirmed small cell lung cancer. Confirmation will be done at each participating site.
2. Have relapsed or progressed after only one prior chemotherapy regimen, which must have been an etoposide-platinum doublet. Eligible patients will be defined as follows:

   "Sensitive" Disease: Patients who had one previous line of chemotherapy and relapsed after > 60 days of completion of treatment.

   "Refractory" Disease: Patients with no response to first-line chemotherapy or progression >60 days after completing treatment.
3. Be ≥ 18 years of age on day of signing informed consent.
4. Have a life expectancy of at least 3 months.
5. Have a performance status of ≤ 1 on the ECOG Performance Scale.
6. Have measurable disease based on RECIST 1.1.
7. Have a tumor tissue specimen available from either a core or excisional biopsy. The tumor specimen should be of adequate size and tumor cellularity to perform whole exome sequencing and immunohistochemistry. In subjects for whom newly obtained samples cannot be obtained (e.g. tumor inaccessible or safety concern), archived tissue may be submitted, if it otherwise satisfies all specimen criteria. Archival samples must have been obtained within 42 days prior to signing consent (please refer to section 12.1 of protocol).
8. Demonstrate adequate organ function as defined in Table 1.

   Table 1. Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥8 g/dL (without transfusion) Renal Serum creatinine

   OR

   Glomerular Filtration Rate (GFR) ≤1.5 X upper limit of normal (ULN)

   OR

   GFR ≥60 mL/min* for patient with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ 1.5 X ULN

   OR

   Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN

   OR

   ≤ 5 X ULN for patients with liver metastases Albumin ≥ 2.5 mg/dL

   *GFR should be calculated per institutional standards.
9. Female patients of childbearing potential should have a negative urine or serum pregnancy within 72 hours of starting treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female patients of childbearing potential must be willing to an adequate method of contraception as outlined in Section 14.4.1 - Contraception for the course of the study through 120 days after the last dose of study medication (see Section 13.4.1). Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male patients must agree to use an adequate method of contraception as outlined in Section 14.4.1 - Contraception - starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* The patient must be excluded from participating in the trial if the patient:

  1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 14 days of the first dose of treatment.
  2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
  3. Has had a prior monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 14 days earlier.
  4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

     Note: Patients with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.
  5. Has undergone major surgery, he/she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
  6. Has a known additional malignancy that is progressing or requires active treatment.
  7. Has known active central nervous system (CNS) metastases. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
  8. Has known carcinomatous meningitis.
  9. Has an active autoimmune disease requiring systemic treatment in the past 2 years or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
  10. Has evidence of interstitial lung disease, or history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
  11. Has an active infection requiring systemic therapy.
  12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
  13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
  15. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
  16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
  17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
  18. Has received a live vaccine within 30 days prior to the planned first dose of study therapy.

      Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
  19. Has a known history of active TB (Bacillus Tuberculosis).
  20. Hypersensitivity to pembrolizumab or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bertagnolli, MD, Principal Investigator — Alliance Foundation Trials; Thomas Stinchcombe, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Metro MN Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Gaspar LE, McNamara EJ, Gay EG, Putnam JB, Crawford J, Herbst RS, Bonner JA. Small-cell lung cancer: prognostic factors and changing treatment over 15 years. Clin Lung Cancer. 2012 Mar;13(2):115-22. doi: 10.1016/j.cllc.2011.05.008. Epub 2011 Oct 14. PMID 22000695
- [Background] Varghese AM, Zakowski MF, Yu HA, Won HH, Riely GJ, Krug LM, Kris MG, Rekhtman N, Ladanyi M, Wang L, Berger MF, Pietanza MC. Small-cell lung cancers in patients who never smoked cigarettes. J Thorac Oncol. 2014 Jun;9(6):892-6. doi: 10.1097/JTO.0000000000000142. PMID 24828667
- [Background] Ou SH, Ziogas A, Zell JA. Prognostic factors for survival in extensive stage small cell lung cancer (ED-SCLC): the importance of smoking history, socioeconomic and marital statuses, and ethnicity. J Thorac Oncol. 2009 Jan;4(1):37-43. doi: 10.1097/JTO.0b013e31819140fb. PMID 19096304
- [Background] Krug LM, Kris MG, Rosenzweig K, Travis W. Small cell and other neuroendocrine tumors of the lung. In: DeVita VT, Hellman S, Rosenberg SA, eds. Cancer: Principles & Practice of Oncolology. 8th ed: Lippincott, Williams, and Wilkins; 2008.
- [Background] von Pawel J, Schiller JH, Shepherd FA, Fields SZ, Kleisbauer JP, Chrysson NG, Stewart DJ, Clark PI, Palmer MC, Depierre A, Carmichael J, Krebs JB, Ross G, Lane SR, Gralla R. Topotecan versus cyclophosphamide, doxorubicin, and vincristine for the treatment of recurrent small-cell lung cancer. J Clin Oncol. 1999 Feb;17(2):658-67. doi: 10.1200/JCO.1999.17.2.658. PMID 10080612
- [Background] Ardizzoni A, Hansen H, Dombernowsky P, Gamucci T, Kaplan S, Postmus P, Giaccone G, Schaefer B, Wanders J, Verweij J. Topotecan, a new active drug in the second-line treatment of small-cell lung cancer: a phase II study in patients with refractory and sensitive disease. The European Organization for Research and Treatment of Cancer Early Clinical Studies Group and New Drug Development Office, and the Lung Cancer Cooperative Group. J Clin Oncol. 1997 May;15(5):2090-6. doi: 10.1200/JCO.1997.15.5.2090. PMID 9164222
- [Background] Eckardt J, Gralla R, Palmer MC, et al. Topotecan as second-line therapy in patients with small cell lung cancer: a phase II study. Ann Oncol 1996;7:107 (abstr 513).
- [Background] Depierre A, von Pawel J, Hans L, et al. Evaluation of Topotecan (Hycamtin) in relapsed small-cell lung cancer (SCLC): A multicenter phase II study. Lung Cancer 1997;18:35 (abstract 126).
- [Background] Eckardt J, Depierre A, Ardizzoni A, von Pawel J, Fields SZ. Pooled analysis of topotecan in the second-line treatment of patients with sensitive small cell lung cancer. Proc Am Soc Clin Oncol 1997;16:452a (abstr 1624).
- [Background] O'Brien M, Eckardt J, Ramlau R. Recent advances with topotecan in the treatment of lung cancer. Oncologist. 2007 Oct;12(10):1194-204. doi: 10.1634/theoncologist.12-10-1194. PMID 17962613
- [Background] Koschel R, Huber RM, Gatzemeier U, et al. Topotecan in Second-Line Treatment of Small Cell Lung Cancer Reduced Toxicity with Individualized Therapy. Lung Cancer 2000;29:42 (abstract 135).
- [Background] Huber RM, Reck M, Gosse H, von Pawel J, Mezger J, Saal JG, Kleinschmidt R, Steppert C, Steppling H. Efficacy of a toxicity-adjusted topotecan therapy in recurrent small cell lung cancer. Eur Respir J. 2006 Jun;27(6):1183-9. doi: 10.1183/09031936.06.00015605. Epub 2006 Feb 15. PMID 16481389
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Sharpe AH, Freeman GJ. The B7-CD28 superfamily. Nat Rev Immunol. 2002 Feb;2(2):116-26. doi: 10.1038/nri727. PMID 11910893
- [Background] Johnson BJ, Costelloe EO, Fitzpatrick DR, Haanen JB, Schumacher TN, Brown LE, Kelso A. Single-cell perforin and granzyme expression reveals the anatomical localization of effector CD8+ T cells in influenza virus-infected mice. Proc Natl Acad Sci U S A. 2003 Mar 4;100(5):2657-62. doi: 10.1073/pnas.0538056100. Epub 2003 Feb 24. PMID 12601154
- [Background] Thompson RH, Dong H, Kwon ED. Implications of B7-H1 expression in clear cell carcinoma of the kidney for prognostication and therapy. Clin Cancer Res. 2007 Jan 15;13(2 Pt 2):709s-715s. doi: 10.1158/1078-0432.CCR-06-1868. PMID 17255298
- [Background] Koyama K, Kagamu H, Miura S, Hiura T, Miyabayashi T, Itoh R, Kuriyama H, Tanaka H, Tanaka J, Yoshizawa H, Nakata K, Gejyo F. Reciprocal CD4+ T-cell balance of effector CD62Llow CD4+ and CD62LhighCD25+ CD4+ regulatory T cells in small cell lung cancer reflects disease stage. Clin Cancer Res. 2008 Nov 1;14(21):6770-9. doi: 10.1158/1078-0432.CCR-08-1156. PMID 18980970
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Terawaki S, Tanaka Y, Nagakura T, Hayashi T, Shibayama S, Muroi K, Okazaki T, Mikami B, Garboczi DN, Honjo T, Minato N. Specific and high-affinity binding of tetramerized PD-L1 extracellular domain to PD-1-expressing cells: possible application to enhance T cell function. Int Immunol. 2007 Jul;19(7):881-90. doi: 10.1093/intimm/dxm059. Epub 2007 Jul 2. PMID 17606978
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Saunders PA, Hendrycks VR, Lidinsky WA, Woods ML. PD-L2:PD-1 involvement in T cell proliferation, cytokine production, and integrin-mediated adhesion. Eur J Immunol. 2005 Dec;35(12):3561-9. doi: 10.1002/eji.200526347. PMID 16278812
- [Background] Robert C, Ribas A, Wolchok JD, Hodi FS, Hamid O, Kefford R, Weber JS, Joshua AM, Hwu WJ, Gangadhar TC, Patnaik A, Dronca R, Zarour H, Joseph RW, Boasberg P, Chmielowski B, Mateus C, Postow MA, Gergich K, Elassaiss-Schaap J, Li XN, Iannone R, Ebbinghaus SW, Kang SP, Daud A. Anti-programmed-death-receptor-1 treatment with pembrolizumab in ipilimumab-refractory advanced melanoma: a randomised dose-comparison cohort of a phase 1 trial. Lancet. 2014 Sep 20;384(9948):1109-17. doi: 10.1016/S0140-6736(14)60958-2. Epub 2014 Jul 15. PMID 25034862
- [Background] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Graus F, Dalmou J, Rene R, Tora M, Malats N, Verschuuren JJ, Cardenal F, Vinolas N, Garcia del Muro J, Vadell C, Mason WP, Rosell R, Posner JB, Real FX. Anti-Hu antibodies in patients with small-cell lung cancer: association with complete response to therapy and improved survival. J Clin Oncol. 1997 Aug;15(8):2866-72. doi: 10.1200/JCO.1997.15.8.2866. PMID 9256130
- [Background] Tanio Y, Watanabe M, Osaki T, Tachibana I, Kawase I, Kuritani T, Saito S, Masuno T, Kodama N, Furuse K, et al. High sensitivity to peripheral blood lymphocytes and low HLA-class I antigen expression of small cell lung cancer cell lines with diverse chemo-radiosensitivity. Jpn J Cancer Res. 1992 Jul;83(7):736-45. doi: 10.1111/j.1349-7006.1992.tb01974.x. PMID 1325431
- [Background] Yazawa T, Kamma H, Fujiwara M, Matsui M, Horiguchi H, Satoh H, Fujimoto M, Yokoyama K, Ogata T. Lack of class II transactivator causes severe deficiency of HLA-DR expression in small cell lung cancer. J Pathol. 1999 Jan;187(2):191-9. doi: 10.1002/(SICI)1096-9896(199901)187:23.0.CO;2-3. PMID 10365094
- [Background] Schultheis AM, Scheel AH, Ozretic L, George J, Thomas RK, Hagemann T, Zander T, Wolf J, Buettner R. PD-L1 expression in small cell neuroendocrine carcinomas. Eur J Cancer. 2015 Feb;51(3):421-6. doi: 10.1016/j.ejca.2014.12.006. Epub 2015 Jan 9. PMID 25582496
- [Background] Lynch TJ, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Neal J, Lu H, Cuillerot JM, Reck M. Ipilimumab in combination with paclitaxel and carboplatin as first-line treatment in stage IIIB/IV non-small-cell lung cancer: results from a randomized, double-blind, multicenter phase II study. J Clin Oncol. 2012 Jun 10;30(17):2046-54. doi: 10.1200/JCO.2011.38.4032. Epub 2012 Apr 30. PMID 22547592
- [Background] Reck M, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Lu H, Cuillerot JM, Lynch TJ. Ipilimumab in combination with paclitaxel and carboplatin as first-line therapy in extensive-disease-small-cell lung cancer: results from a randomized, double-blind, multicenter phase 2 trial. Ann Oncol. 2013 Jan;24(1):75-83. doi: 10.1093/annonc/mds213. Epub 2012 Aug 2. PMID 22858559
- [Background] Ott PA, Elez E, Hiret S, et al. Pembrolizumab for Extensive Stage Disease SCLC: Efficacy and Relationship with PD-L1 Expression. 16th World Conference on Lung Cancer 2015;Abstract 3285.
- [Background] George J, Lim JS, Jang SJ, Cun Y, Ozretic L, Kong G, Leenders F, Lu X, Fernandez-Cuesta L, Bosco G, Muller C, Dahmen I, Jahchan NS, Park KS, Yang D, Karnezis AN, Vaka D, Torres A, Wang MS, Korbel JO, Menon R, Chun SM, Kim D, Wilkerson M, Hayes N, Engelmann D, Putzer B, Bos M, Michels S, Vlasic I, Seidel D, Pinther B, Schaub P, Becker C, Altmuller J, Yokota J, Kohno T, Iwakawa R, Tsuta K, Noguchi M, Muley T, Hoffmann H, Schnabel PA, Petersen I, Chen Y, Soltermann A, Tischler V, Choi CM, Kim YH, Massion PP, Zou Y, Jovanovic D, Kontic M, Wright GM, Russell PA, Solomon B, Koch I, Lindner M, Muscarella LA, la Torre A, Field JK, Jakopovic M, Knezevic J, Castanos-Velez E, Roz L, Pastorino U, Brustugun OT, Lund-Iversen M, Thunnissen E, Kohler J, Schuler M, Botling J, Sandelin M, Sanchez-Cespedes M, Salvesen HB, Achter V, Lang U, Bogus M, Schneider PM, Zander T, Ansen S, Hallek M, Wolf J, Vingron M, Yatabe Y, Travis WD, Nurnberg P, Reinhardt C, Perner S, Heukamp L, Buttner R, Haas SA, Brambilla E, Peifer M, Sage J, Thomas RK. Comprehensive genomic profiles of small cell lung cancer. Nature. 2015 Aug 6;524(7563):47-53. doi: 10.1038/nature14664. Epub 2015 Jul 13. PMID 26168399
- [Background] Pleasance ED, Stephens PJ, O'Meara S, McBride DJ, Meynert A, Jones D, Lin ML, Beare D, Lau KW, Greenman C, Varela I, Nik-Zainal S, Davies HR, Ordonez GR, Mudie LJ, Latimer C, Edkins S, Stebbings L, Chen L, Jia M, Leroy C, Marshall J, Menzies A, Butler A, Teague JW, Mangion J, Sun YA, McLaughlin SF, Peckham HE, Tsung EF, Costa GL, Lee CC, Minna JD, Gazdar A, Birney E, Rhodes MD, McKernan KJ, Stratton MR, Futreal PA, Campbell PJ. A small-cell lung cancer genome with complex signatures of tobacco exposure. Nature. 2010 Jan 14;463(7278):184-90. doi: 10.1038/nature08629. Epub 2009 Dec 16. PMID 20016488
- [Background] Rudin CM, Durinck S, Stawiski EW, Poirier JT, Modrusan Z, Shames DS, Bergbower EA, Guan Y, Shin J, Guillory J, Rivers CS, Foo CK, Bhatt D, Stinson J, Gnad F, Haverty PM, Gentleman R, Chaudhuri S, Janakiraman V, Jaiswal BS, Parikh C, Yuan W, Zhang Z, Koeppen H, Wu TD, Stern HM, Yauch RL, Huffman KE, Paskulin DD, Illei PB, Varella-Garcia M, Gazdar AF, de Sauvage FJ, Bourgon R, Minna JD, Brock MV, Seshagiri S. Comprehensive genomic analysis identifies SOX2 as a frequently amplified gene in small-cell lung cancer. Nat Genet. 2012 Oct;44(10):1111-6. doi: 10.1038/ng.2405. Epub 2012 Sep 2. PMID 22941189
- [Background] Peifer M, Fernandez-Cuesta L, Sos ML, George J, Seidel D, Kasper LH, Plenker D, Leenders F, Sun R, Zander T, Menon R, Koker M, Dahmen I, Muller C, Di Cerbo V, Schildhaus HU, Altmuller J, Baessmann I, Becker C, de Wilde B, Vandesompele J, Bohm D, Ansen S, Gabler F, Wilkening I, Heynck S, Heuckmann JM, Lu X, Carter SL, Cibulskis K, Banerji S, Getz G, Park KS, Rauh D, Grutter C, Fischer M, Pasqualucci L, Wright G, Wainer Z, Russell P, Petersen I, Chen Y, Stoelben E, Ludwig C, Schnabel P, Hoffmann H, Muley T, Brockmann M, Engel-Riedel W, Muscarella LA, Fazio VM, Groen H, Timens W, Sietsma H, Thunnissen E, Smit E, Heideman DA, Snijders PJ, Cappuzzo F, Ligorio C, Damiani S, Field J, Solberg S, Brustugun OT, Lund-Iversen M, Sanger J, Clement JH, Soltermann A, Moch H, Weder W, Solomon B, Soria JC, Validire P, Besse B, Brambilla E, Brambilla C, Lantuejoul S, Lorimier P, Schneider PM, Hallek M, Pao W, Meyerson M, Sage J, Shendure J, Schneider R, Buttner R, Wolf J, Nurnberg P, Perner S, Heukamp LC, Brindle PK, Haas S, Thomas RK. Integrative genome analyses identify key somatic driver mutations of small-cell lung cancer. Nat Genet. 2012 Oct;44(10):1104-10. doi: 10.1038/ng.2396. Epub 2012 Sep 2. PMID 22941188
- [Background] Lawrence MS, Stojanov P, Polak P, Kryukov GV, Cibulskis K, Sivachenko A, Carter SL, Stewart C, Mermel CH, Roberts SA, Kiezun A, Hammerman PS, McKenna A, Drier Y, Zou L, Ramos AH, Pugh TJ, Stransky N, Helman E, Kim J, Sougnez C, Ambrogio L, Nickerson E, Shefler E, Cortes ML, Auclair D, Saksena G, Voet D, Noble M, DiCara D, Lin P, Lichtenstein L, Heiman DI, Fennell T, Imielinski M, Hernandez B, Hodis E, Baca S, Dulak AM, Lohr J, Landau DA, Wu CJ, Melendez-Zajgla J, Hidalgo-Miranda A, Koren A, McCarroll SA, Mora J, Crompton B, Onofrio R, Parkin M, Winckler W, Ardlie K, Gabriel SB, Roberts CWM, Biegel JA, Stegmaier K, Bass AJ, Garraway LA, Meyerson M, Golub TR, Gordenin DA, Sunyaev S, Lander ES, Getz G. Mutational heterogeneity in cancer and the search for new cancer-associated genes. Nature. 2013 Jul 11;499(7457):214-218. doi: 10.1038/nature12213. Epub 2013 Jun 16. PMID 23770567
- [Background] Snyder A, Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, Walsh LA, Postow MA, Wong P, Ho TS, Hollmann TJ, Bruggeman C, Kannan K, Li Y, Elipenahli C, Liu C, Harbison CT, Wang L, Ribas A, Wolchok JD, Chan TA. Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med. 2014 Dec 4;371(23):2189-2199. doi: 10.1056/NEJMoa1406498. Epub 2014 Nov 19. PMID 25409260
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Eckardt JR, von Pawel J, Pujol JL, Papai Z, Quoix E, Ardizzoni A, Poulin R, Preston AJ, Dane G, Ross G. Phase III study of oral compared with intravenous topotecan as second-line therapy in small-cell lung cancer. J Clin Oncol. 2007 May 20;25(15):2086-92. doi: 10.1200/JCO.2006.08.3998. PMID 17513814
- [Background] J-C S, O F, L H, et al. LATE BREAKING ABSTRACT: Efficacy and Safety of Pembrolizumab (Pembro; MK-3475) for Patients (Pts) With Previously Treated Advanced Non-Small Cell Lung Cancer (NSCLC) Enrolled in KEYNOTE-001. European Society of Medical Oncology Annual Meeting 2015:33LBA.
- [Background] Hellmann M, Creelan B, Woo K, et al. Smoking history and response to nivolumab in patients with advanced NSCLCs. Ann Oncol 2014;25.
- [Background] Matsushita H, Vesely MD, Koboldt DC, Rickert CG, Uppaluri R, Magrini VJ, Arthur CD, White JM, Chen YS, Shea LK, Hundal J, Wendl MC, Demeter R, Wylie T, Allison JP, Smyth MJ, Old LJ, Mardis ER, Schreiber RD. Cancer exome analysis reveals a T-cell-dependent mechanism of cancer immunoediting. Nature. 2012 Feb 8;482(7385):400-4. doi: 10.1038/nature10755. PMID 22318521
- [Background] Castle JC, Kreiter S, Diekmann J, Lower M, van de Roemer N, de Graaf J, Selmi A, Diken M, Boegel S, Paret C, Koslowski M, Kuhn AN, Britten CM, Huber C, Tureci O, Sahin U. Exploiting the mutanome for tumor vaccination. Cancer Res. 2012 Mar 1;72(5):1081-91. doi: 10.1158/0008-5472.CAN-11-3722. Epub 2012 Jan 11. PMID 22237626
- [Background] Lennerz V, Fatho M, Gentilini C, Frye RA, Lifke A, Ferel D, Wolfel C, Huber C, Wolfel T. The response of autologous T cells to a human melanoma is dominated by mutated neoantigens. Proc Natl Acad Sci U S A. 2005 Nov 1;102(44):16013-8. doi: 10.1073/pnas.0500090102. Epub 2005 Oct 24. PMID 16247014
- [Background] van Rooij N, van Buuren MM, Philips D, Velds A, Toebes M, Heemskerk B, van Dijk LJ, Behjati S, Hilkmann H, El Atmioui D, Nieuwland M, Stratton MR, Kerkhoven RM, Kesmir C, Haanen JB, Kvistborg P, Schumacher TN. Tumor exome analysis reveals neoantigen-specific T-cell reactivity in an ipilimumab-responsive melanoma. J Clin Oncol. 2013 Nov 10;31(32):e439-42. doi: 10.1200/JCO.2012.47.7521. Epub 2013 Sep 16. No abstract available. PMID 24043743
- [Background] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- [Background] Engels B, Engelhard VH, Sidney J, Sette A, Binder DC, Liu RB, Kranz DM, Meredith SC, Rowley DA, Schreiber H. Relapse or eradication of cancer is predicted by peptide-major histocompatibility complex affinity. Cancer Cell. 2013 Apr 15;23(4):516-26. doi: 10.1016/j.ccr.2013.03.018. PMID 23597565
- [Background] Lundegaard C, Lund O, Nielsen M. Accurate approximation method for prediction of class I MHC affinities for peptides of length 8, 10 and 11 using prediction tools trained on 9mers. Bioinformatics. 2008 Jun 1;24(11):1397-8. doi: 10.1093/bioinformatics/btn128. Epub 2008 Apr 14. PMID 18413329
- [Background] Lundegaard C, Lamberth K, Harndahl M, Buus S, Lund O, Nielsen M. NetMHC-3.0: accurate web accessible predictions of human, mouse and monkey MHC class I affinities for peptides of length 8-11. Nucleic Acids Res. 2008 Jul 1;36(Web Server issue):W509-12. doi: 10.1093/nar/gkn202. Epub 2008 May 7. PMID 18463140
- [Background] Andersen RS, Kvistborg P, Frosig TM, Pedersen NW, Lyngaa R, Bakker AH, Shu CJ, Straten Pt, Schumacher TN, Hadrup SR. Parallel detection of antigen-specific T cell responses by combinatorial encoding of MHC multimers. Nat Protoc. 2012 Apr 12;7(5):891-902. doi: 10.1038/nprot.2012.037. PMID 22498709
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Fleming TR and Harrington DP. (1991). Counting Processes and Survival Analysis. New York, NY: John Wiley & Sons.

RESULTS

PARTICIPANT FLOW:
Groups:
- Topotecan (Arm A): Topotecan IV at 1.25 mg/m2 Days 1-5 of every 21 day cycle.
- Pembrolizumab (Arm B): Pembrolizumab IV 200mg infusion Day 1 of every 21 day cycle.
Period: Non-cross Over Phase
Arm/Group | Topotecan (Arm A) | Pembrolizumab (Arm B)
Started | 3 | 6
Completed | 2 | 6
Not Completed | 1 | 0
Not completed — Patient deterioration before starting protocol treatment | 1 | 0
Period: Cross Over Phase
Arm/Group | Topotecan (Arm A) | Pembrolizumab (Arm B)
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Topotecan: Topotecan IV at 1.25 mg/m2 Days 1-5 of every 21 day cycle.
- Crossover: Topotecan IV at 1.25 mg/m2 Days 1-5 of every 21 day cycle. Then at progression of disease by RECIST 1.1. Patients then receive pembrolizumab 200 mg IV every 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Topotecan | Pembrolizumab | Crossover | Total
Number analyzed (Participants) | 1 | 6 | 2 | 9
Age, Continuous [Median (Full Range); unit: years] | 82 [82 to 82] | 71 [55 to 75] | 63.5 [63 to 64] | 69 [55 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 7
  Male | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 6 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 1 | 6 | 1 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: This phase II study will determine if there is a benefit in progression free survival (PFS) for SCLC patients receiving pembrolizumab (Experimental arm) as compared to topotecan (Control arm) in the second-line settingSCLC patients receiving pembrolizumab (Experimental arm) as compared to topotecan (Control arm) in the second-line setting. RECIST Version 1.1 was used in this study for assessment for tumor response. Progression (PD): At least one of the following must be true: a. At least one new malignant lesion, which also includes any lymph node that was normal at baseline (< 1.0 cm short axis) and increased to ≥ 1.0 cm short axis during follow-up. b. At least a 20% increase in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the MSD. In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD.
Time Frame: 4.2 months
Population: All patients that were treated and evaluated for disease. Crossover patients were analyzed using their time on Arm A.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Topotecan (Arm A + Crossover Patients): Topotecan IV at 1.25 mg/m2 Days 1-5 of every 21 day cycle.
Arm/Group | Topotecan (Arm A + Crossover Patients) | Pembrolizumab
Number analyzed (Participants) | 2 | 6
Months | 1.4 [NA to NA] — Insufficient number of participants with events below the level of detection to determine the lower and upper limits of the Confidence Intervals. | 1.5 [1.1 to NA] — insufficient number of participants with events below the level of detection to determine the upper limits of the Confidence Intervals

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival will be calculated from the time a patient is registered until the time of death or discontinuation of followup
Time Frame: 20 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Topotecan (Arm A) | Pembrolizumab (Arm B)
Number analyzed (Participants) | 2 | 6
Months | NA [3.1 to NA] — Not enough events to calculate median or upper limit | 10.7 [3.6 to NA] — Not enough events to calculate upper limit

3. Secondary Outcome: Overall Response Percentage
Description: RECIST Version 1.1* will be used in this study for assessment for tumor response.
  Complete Response (CR): All of the following must be true:
  1. Disappearance of all target lesions.
  2. Each target lymph node must have reduction in short axis to < 1.0 cm. • Partial Response (PR): At least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the BSD
Time Frame: 4.2 months
Measure: Number; unit: percentage of participants
Arm/Group | Topotecan (Arm A) | Pembrolizumab (Arm B)
Number analyzed (Participants) | 2 | 6
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 20 months
Description: The crossover arm consists of two of the Arm A patients after they progressed and chose to cross to Arm B treatment.
Arm/Group | Topotecan | Pembrolizumab | Crossover
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/6 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/6 | 2/2
Other Adverse Events (participants affected / at risk) | 2/3 | 5/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topotecan (N=3) | Pembrolizumab (N=6) | Crossover (N=2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topotecan (N=3) | Pembrolizumab (N=6) | Crossover (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 2 (7) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (2) | 2 (4)
White blood cell decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT02963090/Prot_SAP_001.pdf